CLINICAL TRIAL: NCT04841837
Title: Effect of Time-restricted Eating on Blood Glucose and Behavior in Patients With Type 2 Diabetes Mellitus
Acronym: TREAT BB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006761-M2021024
Record Dates: First submitted 2021-04-06; First posted 2021-04-12 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Time-restricted feeding; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-restricted feeding (Experimental): Restrict all calorie intake within a self-selected 10-hours window for 12 weeks, without necessarily altering diet quality and quantity
  Interventions: Behavioral: Time-restricted feeding

INTERVENTIONS:
Behavioral: Time-restricted feeding — limit daily food intake to a period of 10 hours

SUMMARY:
Diet management could improve blood and weight control in patients with diabetes mellitus. Time-restricted feeding is a novel dietary tool that limits time of energy intake without altering diet quality or quantity. This study aims to assess the effect of 10-hour time-restricted feeding on metabolism and behavior in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes mellitus
2. HbA1c 7.0% to 8.5%
3. BMI ≥ 24 kg/m2
4. Time of energy intake ≥ 12 hours per day, ≥ 4 days per week
5. Ability to use smart phone and app, to follow study protocol
6. Sign informed consent

Exclusion Criteria:

1. Use insulin, long-acting insulin secretagogues, GLP-1 receptor agonist, DPP-4 inhibitor, SGLT-2 inhibitor
2. Suffer from disease influence eating: mental disease, subtotal gastrectomy, inflammatory bowel disease, uncontrolled thyroid disease
3. Work state affect eating time: constant night duty, constant long-haul international travel
4. Smoking
5. Drinking
6. Severe disease: severe cardiovascular and cerebrovascular disease, uncontrolled arrhythmia, heart failure, acute and chronic renal dysfunction, liver cirrhosis, malignancy, anemia
7. Suffered from infectious disease: pulmonary tuberculosis, AIDS
8. Dyskinesia
9. Body weight change ≥ 5 kg in the past 3 months
10. Hospitalized in the past 3 months
11. Used antibiotics for ≥ 3 days in the past 3 months
12. Diagnosed with type 1 diabetes mellitus
13. Pregnancy, lactating
14. Participating in other clinical trials in the past 1 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | through study completion, an average of 12 weeks
Mean blood glucose | through study completion, an average of 12 weeks
Time in range | through study completion, an average of 12 weeks

SECONDARY OUTCOMES:
Compliance of time-restricted feeding | through study completion, an average of 12 weeks
  Percent of days when the participants follow 10-hours window of calorie intake
Adverse event | through study completion, an average of 12 weeks
type and proportion of intestinal flora | through study completion, an average of 12 weeks
  Collect fecal specimens, analyze the types and proportion of intestinal flora
Body weight (kg) | through study completion, an average of 12 weeks
  Electronic weighing scale will be used to weigh participants
Body composition (fat and muscle mass) | through study completion, an average of 12 weeks
  Body composition analyzer will be used to analyze fat and muscle mass

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No